CLINICAL TRIAL: NCT02488824
Title: Effect of Heat Exposure on Cognition in Persons With Higher Cord Lesions
Brief Title: Effect of Heat Exposure on Cognition in Persons With Tetraplegia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: D1734-P; HAN-15-013 (Other: James J. Peters Veterans Affairs Medical Center); 01613 (Other: James J Peters VAMC IRB)
Record Dates: First submitted 2015-04-20; First posted 2015-07-02 (Estimated); Results first posted 2019-11-01 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Tetraplegia; Hypothermia; Mild Cognitive Impairment
Keywords: Quadriplegia; Paraplegia; Spinal Cord Injury; Body Temperature Regulation; Mild Cognitive Impairment
MeSH Terms: conditions — Quadriplegia; Hypothermia; Cognitive Dysfunction; Paraplegia; Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Warm Temperature Exposure in Tetraplegia (Experimental): Subjects are persons with higher-level spinal cord injury, levels C3 to T4, and ASIA Impairment Scale (AIS) level A and B, ages 18-68 years. Procedure is exposure to warm temperature (95 degrees Fahrenheit) for up to 2 hours in a temperature-controlled room in order to assess the body's temperature-regulating mechanisms and any associated change in cognitive performance
  Interventions: Procedure: Warm Temperature
- Warm Temperature Exposure in Able-Bodied (Active Comparator): Subjects are able-bodied controls matched with participants with tetraplegia for age and gender. Procedure is exposure to warm temperature (95 degrees Fahrenheit) for up to 2 hours in a temperature-controlled room in order to assess the body's temperature-regulating mechanisms and any associated change in cognitive performance
  Interventions: Procedure: Warm Temperature

INTERVENTIONS:
Procedure: Warm Temperature — Subjects will be exposed to a routinely encountered warm temperature (95 F) for up to to 2 hours, depending on their vital signs (BP, HR, Tcore) and tolerance (comfort).
  Other Names: 95 F

SUMMARY:
The ability to maintain normal body temperature (Tcore) is impaired in persons with tetraplegia: subnormal Tcore and vulnerability to hypothermia (<95 F) have been documented in this population after exposure to even mild environmental temperatures. However, no work to date has addressed the effect of subnormal Tcore on cognitive performance in persons with tetraplegia despite studies with able-bodied (AB) individuals that have documented progressive decline in various aspects of cognitive performance associated with the magnitude of the depression in Tcore. The investigators' study will confirm and extend their initial observations in persons with higher cord lesions who have subnormal Tcore to show that cognitive performance will be improved by raising Tcore to euthermic levels. This improvement should be associated with greater function and independence, reintegration into society, and an improved quality of life.

Specific Aims: During exposure to 95 F for up to 120 minutes in the seated position, the investigators' aims are:

Primary Specific Aim: To determine if a modest rise in Tcore to euthermic levels has a positive effect on cognitive performance (attention, working memory, processing speed, and executive function) in persons with higher-level spinal cord injury (SCI).

Primary Hypothesis: Based on the investigators' pilot data: (1) 80% of persons with SCI will demonstrate an increase of 1 F in Tcore, while none of the AB controls will demonstrate such an increase; (2) 80% of persons with SCI will have an improvement of at least one T-score in Stroop Interference scores (a validated measure of executive function), while none of the AB controls will demonstrate a change in cognitive performance.

Secondary Specific Aim: To determine changes in: (1) The average of distal skin temperatures; (2) Sweat rate; and (3) Subjective rating of thermal sensitivity.

Secondary Hypothesis: Persons with SCI will have less of a percent change in average distal skin temperatures and sweat rate, and will report blunted ratings of thermal sensitivity compared to that of AB controls.

DETAILED DESCRIPTION:
This study will investigate the physiological and cognitive responses to warm exposure in persons with SCI who have subnormal Tcore and in AB persons who are euthermic. The positive effect that an increase in Tcore will be expected to have on cognitive performance, specifically working memory and executive function, will be demonstrated. These two areas of cognitive performance are vital for the ability to optimally care for one's self, at which persons with higher cord lesions must excel in order to ensure health, and for the ability to attain the maximal degree of independence possible.

Preparation for Study Visits: Subjects will be instructed to avoid caffeine and alcohol, maintain normal salt and water intake, and avoid strenuous exercise for 24 hours prior to the study. Subjects will be asked to eat a light, standard meal (plain bagel or 2 pieces of toast) 2 hours prior to their visit. Subjects will be asked to empty their bladders prior to their visit and again upon arrival, if needed. Subjects will wear minimal clothing during the study to maximize skin exposure to the warm temperature.

Instrumentation: Subjects with SCI will be asked to remain in their wheelchairs and AB controls will be placed in a manual wheelchair where they will remain seated and relatively still for the duration of the study visit. A thin, flexible rectal sensor will be placed 4 inches beyond the anal sphincter for Tcore collection, and skin sensors will be secured at 15 sites above and below the level of lesion for collection of skin temperature (Tsk). Sweat collection capsules will be placed on the left bicep, the left forearm, the left thigh and the left calf for measurement of sweat rate by QSweat methodology (QS). Laser Doppler flowmetry will be used to measure changes in microvascular perfusion (MVP) by placing a Doppler probe on the back of both hands and both feet to confirm peripheral blood vessel dilation. An automated blood pressure cuff will be placed above the left elbow to measure brachial BP.

Baseline Collection (BL): At the end of a 30-minute acclimation period at 81 F, a baseline collection of the following parameters will be performed for 15 minutes: Tcore and Tsk will be continuously monitored; BP, heart rate (HR), and thermal sensitivity (TS) will be measured in 10-minute intervals; and MVP and QS will be measured in 15-minute intervals. After 15 minutes, a battery of cognitive tests will be administered to establish baseline cognitive performance.

Thermal Challenge (Heat): Following completion of the BL period, subjects will be wheeled into a pre-heated (95 F) thermal chamber for up to 120 minutes or until Tcore increases 1 F. Tcore and Tsk will be continuously monitored to ensure subjects' safety throughout the protocol, while HR, BP, and TS will be assessed at 10-minute intervals. MVP and QS will be measured every 30 minutes. The battery of cognitive tests utilized during BL collection will be administered when Tcore increases 1 F from BL values (for subjects with tetraplegia) or after 100 minutes (for controls) to determine any change in cognition after exposure to 95 F. An increase in Tcore 1 F, significant changes in BP, or subject discomfort will result in termination of the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Duration of injury 1 year
* Level of SCI C3-T4, AIS A & B
* Tcore at BL <98.6 F (subnormal core body temperature)
* Euhydration
* Gender and age-matched ( 5 years) AB controls (between 18-68 years of age)

Exclusion Criteria:

* Known heart, kidney, peripheral vascular, or cerebral vascular disease
* High blood pressure
* History of traumatic brain injury or diagnosed cognitive impairment
* Untreated thyroid disease
* Diabetes mellitus
* Acute illness or infection
* Dehydration
* Smoking
* Pregnancy
* Broken, inflamed, or otherwise fragile skin

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2018-09-04 (Actual); Study Completion 2018-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Philip Handrakis, PT DPT EdD, Principal Investigator — James J. Peters Veterans Affairs Medical Center
Locations (1):
- James J. Peters VA Medical Center, Bronx, NY, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Click here for more information about this study: Effect of Heat Exposure on Cognition in Persons with Higher Cord Lesions — http://scirc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Warm Temperature Exposure in Tetraplegia: Subjects are persons with higher-level spinal cord injury, levels C3 to T4, and ASIA Impairment Scale (AIS) level A and B, ages 18-68 years. Procedure is exposure to warm temperature (95 deg F) for up to 2 hours in a temperature-controlled room in order to assess the body's temperature-regulating mechanisms and any associated change in cognitive performance
  Warm Temperature: Subjects will be exposed to a routinely encountered warm temperature (95 deg F) for up to to 2 hours, depending on their vital signs (BP, HR, Tcore) and tolerance (comfort).
- Active Comparator: Warm Temperature Exposure in Able-Bodied: Subjects are able-bodied controls matched with participants with tetraplegia for age and gender. Procedure is exposure to warm temperature (95 deg F) for up to 2 hours in a temperature-controlled room in order to assess the body's temperature-regulating mechanisms and any associated change in cognitive performance
  Warm Temperature: Subjects will be exposed to a routinely encountered warm temperature (95 deg F) for up to to 2 hours, depending on their vital signs (BP, HR, Tcore) and tolerance (comfort).
Period: Overall Study
Arm/Group | Experimental: Warm Temperature Exposure in Tetraplegia | Active Comparator: Warm Temperature Exposure in Able-Bodied
Started | 21 | 20
Completed | 20 | 19
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Experimental: Warm Temperature Exposure in Tetraplegia: Subjects are persons with higher-level spinal cord injury, levels C3 to T4, and ASIA Impairment Scale (AIS) level A and B, ages 18-68 years. Procedure is exposure to warm temperature (95 F) for up to 2 hours in a temperature-controlled room in order to assess the body's temperature-regulating mechanisms and any associated change in cognitive performance
  Warm Temperature: Subjects will be exposed to a routinely encountered warm temperature (95 F) for up to to 2 hours, depending on their vital signs (BP, HR, Tcore) and tolerance (comfort).
- Active Comparator: Warm Temperature Exposure in Able-Bodied: Subjects are able-bodied controls matched with participants with tetraplegia for age and gender. Procedure is exposure to warm temperature (95 F) for up to 2 hours in a temperature-controlled room in order to assess the body's temperature-regulating mechanisms and any associated change in cognitive performance
  Warm Temperature: Subjects will be exposed to a routinely encountered warm temperature (95 F) for up to to 2 hours, depending on their vital signs (BP, HR, Tcore) and tolerance (comfort).
- Total: Total of all reporting groups
Arm/Group | Experimental: Warm Temperature Exposure in Tetraplegia | Active Comparator: Warm Temperature Exposure in Able-Bodied | Total
Number analyzed (Participants) | 20 | 19 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] — Age (in years) of subject
  years | 42.4 (11.4) | 44.3 (13.8) | 43.3 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 16 | 16 | 32
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 4 | 2 | 6
  Black or African American | 1 | 9 | 10
  White | 8 | 6 | 14
  Hispanic or Latino | 7 | 2 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 19 | 39

OUTCOME MEASURES:

1. Primary Outcome: Change in Core Body Temperature From Baseline to 120 Minutes Post Warm Challenge
Description: The investigators measured the effects of warm temperature (95 F) exposure, of up to 120 minutes, on the ability to maintain a constant body temperature (e.g., core temperature of 98.6 F) in both groups of subjects. Core temperature was measured at baseline (thermoneutral) and after 120 minutes of warm temperature exposure (Warm Challenge). The change in core temperature from baseline to 120 minutes of Warm Challenge was calculated.
Time Frame: From Baseline to 120 Minutes
Measure: Mean (Standard Deviation); unit: degrees Centigrade
Arm/Group | Experimental: Warm Temperature Exposure in Tetraplegia | Active Comparator: Warm Temperature Exposure in Able-Bodied
Number analyzed (Participants) | 20 | 19
degrees Centigrade | 0.59 (0.33) | -0.05 (0.23)

2. Primary Outcome: Change in Cognitive Performance From Baseline to 120 Minutes Post Warm Challenge
Description: Cognitive performance was assessed using a neuropsychological battery. Cognitive performance was assessed at 2 time points, at the end of baseline and after heat exposure (warm challenge) in both groups of subjects.
  The Stroop Word test measures processing speed. A T-Score of 50 means "0" difference of actual - predicted score (based on subject's age & education level). T-Scores <40 are considered "low"; T-Scores >40 are considered "normal". Changes of 10 or greater are considered clinically significant. The lowest possible T-Score is 21; the highest possible T-Score is 80.
  The WAIS-IV Digit Span Sequencing measures auditory processing and working memory. Each test score is converted to a scaled score (M=10, SD=3) with higher scores considered better performance. The lowest possible scaled score is 1; the highest possible scaled score is 19.
Time Frame: From Baseline to 120 Minutes
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Experimental: Warm Temperature Exposure in Tetraplegia | Active Comparator: Warm Temperature Exposure in Able-Bodied
Number analyzed (Participants) | 20 | 19
Scores on a scale
  Stroop Word | 6.2 (5.5) | 2.1 (5.4)
  WAIS-IV Digit Span Sequencing | 1.6 (2.1) | 0.3 (2.1)

3. Secondary Outcome: Change in Distal Skin Temperatures From Baseline to 120 Minutes Post Warm Challenge
Description: The investigators measured the effects of warm temperature (95 F) exposure, of up to 120 minutes, on the change in distal skin temperatures in the seated position.
Time Frame: From Baseline to 120 Minutes
Measure: Mean (Standard Deviation); unit: degrees Centigrade
Arm/Group | Experimental: Warm Temperature Exposure in Tetraplegia | Active Comparator: Warm Temperature Exposure in Able-Bodied
Number analyzed (Participants) | 20 | 19
degrees Centigrade | 3.9 (1.7) | 3.9 (2.1)

4. Secondary Outcome: Change in Sweat Rate From Baseline to 120 Minutes Post Warm Challenge
Description: The investigators measured the effects of warm temperature (95 F) exposure, of up to 120 minutes, on the change in sweat rate in the seated position.
Time Frame: From Baseline to 120 Minutes
Measure: Mean (Standard Deviation); unit: nL/min
Arm/Group | Experimental: Warm Temperature Exposure in Tetraplegia | Active Comparator: Warm Temperature Exposure in Able-Bodied
Number analyzed (Participants) | 20 | 19
nL/min | 24.9 (31.8) | 77.0 (52.5)

5. Secondary Outcome: Change in Thermal Sensitivity From Baseline to 120 Minutes Post Warm Challenge
Description: The investigators measured the effects of warm temperature (95 F) exposure, of up to 120 minutes, on the change in thermal sensitivity in the seated position on the 9-Point Thermal sensation scale (+4=very hot, +3=hot, +2=warm, +1=slightly warm, 0=neutral, -1=slightly cool, -2=cool, -3=cold, -4=very cold). A higher score means the subject feels hotter, which, for the identical heat challenge, means less effective thermoregulation.
Time Frame: From Baseline to 120 Minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: Warm Temperature Exposure in Tetraplegia | Active Comparator: Warm Temperature Exposure in Able-Bodied
Number analyzed (Participants) | 20 | 19
score on a scale | 3.3 (1.2) | 2.6 (1.5)

ADVERSE EVENTS:
Time Frame: 3 hours
Description: 1 person with in the group with SCI (Experimental) developed autonomic dysreflexia. 1 person in the able-bodied group (Active comparator) complained of dizziness most likely due to dehydration. The study was stopped for both persons and both persons returned to their baseline status before leaving the lab.
Arm/Group | Experimental: Warm Temperature Exposure in Tetraplegia | Active Comparator: Warm Temperature Exposure in Able-Bodied
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 1/20 | 1/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Warm Temperature Exposure in Tetraplegia (N=20) | Active Comparator: Warm Temperature Exposure in Able-Bodied (N=19)
Autonomic dysreflexia (Vascular disorders) | 1 (1) | 0 (0)
Dehydration (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-09-09): https://cdn.clinicaltrials.gov/large-docs/24/NCT02488824/Prot_SAP_000.pdf